CLINICAL TRIAL: NCT01389726
Title: Comparing Interventions To Improve The Well-Being Of Custodial Grandfamilies
Acronym: COPE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kent State University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Gregory Smith, Ed.D.; Professor, Kent State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: R01NR012256 (NIH); R01NR012256 (NIH)
Record Dates: First submitted 2011-07-05; First posted 2011-07-08 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-08

CONDITIONS: Custodial Grandparents
Keywords: custodial grandparents; kinship caregivers; grandparents raising grandchildren; grandmothers; grandchildren; psychological well-being
MeSH Terms: conditions — Psychological Well-Being | interventions — (tris(diphenylphosphinomethyl)phenylborate)(p-tolylnitrido)iron(I); Cognitive Behavioral Therapy; Self-Help Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Behavioral Parenting Training (Experimental): Triple-P Parenting Training Program (group level)
  Interventions: Behavioral: Behavioral Parent Training
- Cognitive Behavioral Therapy (Experimental): CBT group-level intervention (Designed by Larry Thompson & Dolores Gallagher Thompson)
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Psychosocial-Informational Support (Active Comparator): Standard of Care informational support group
  Interventions: Behavioral: Psychosocial-Informational support

INTERVENTIONS:
Behavioral: Behavioral Parent Training — Triple-P program involves 11 weeks of ongoing group support with contact one time per week with trained group leaders
  Other Names: Triple-P; BPT
  Arms: Behavioral Parenting Training
Behavioral: Cognitive Behavioral Therapy — Support group based intervention involving sessions one time per week for 11 weeks with 9-12 grandmothers, 1 trained professional group leader, and 1 trained peer leader
  Other Names: CBT; Cognitive therapy; Larry Thompson; Dolores Gallagher-Thompson
  Arms: Cognitive Behavioral Therapy
Behavioral: Psychosocial-Informational support — Standard of care normally provided to custodial grandparents. Involves providing information and support in the context of a weekly group meeting with 9-12 grandparents, 1 professional group leader & 1 peer leader over the course of 11 weeks.
  Other Names: Support group
  Arms: Psychosocial-Informational Support

SUMMARY:
This study is a multi-site, four-year long clinical trial study in which several mental health interventions will be delivered to custodial grandmothers and then compared. The study will examine effects on the mental health of these grandmothers and the grandchildren they provide full-time care to in complete absence of the grandchild's birth parents. Grandparents from diverse racial, ethnic, and socio-economic backgrounds will be recruited to test for cultural differences in response to these interventions. This study is important because there is growing evidence that custodial grandchildren are at-risk for psychological difficulties due to neglect and abuse by birth parents, challenges to parenting faced by custodial grandparents, and limited access to needed services. This study is funded by the National Institute of Nursing Research, a division of the National Institutes of Health, and it is anticipated that more than 500 custodial grandfamilies in four sites across the United States will partake.

DETAILED DESCRIPTION:
Although prior studies reveal that custodial grandmothers (CGM) and grandchildren (CGC) face high risk for psychological difficulties, virtually no rigorous studies of psychosocial interventions based on solid conceptual frameworks have been conducted with these vulnerable families. In view of preliminary findings that disrupted parenting mediates the relationship between CGM's psychological distress in the caregiver role and CGC's emotional and behavioral problems, this project involves a randomized clinical trial (RCT) of the comparative feasibility and efficacy of two evidenced-based psychoeducational interventions widely used with other caregiver populations. Grandmothers (N = 504) of CGC (age 5 - 12) will be randomly assigned to one of three conditions: Behavioral Parent Training (BPT; derived from Project KEEP for foster parents; Cognitive Behavioral Therapy (CBT; derived from Coping with Caregiving for caregivers of frail elders); Minimal Support Condition (to control for non-specific treatment factors). The proposed universal interventions include prevention and remediation objectives and involve a group format approach with mental health professionals and grandparent peers serving as co-leaders. The RCT will occur in multiple locations across the US to ensure that findings generalize beyond a single area and that equal numbers of Black (n = 168), Hispanic (n = 168), and White (n = 168) families participate. Prior to the RCT, focus groups will be held separately with CGMs of each race (n = 10 apiece) and experienced practitioners (n = 10) with the aim of assessing the perceived importance and acceptability of recruitment methods, treatment goals, and procedures, including possible differences by race/ethnicity. Multiple-informant and multiple-method assessments during the RCT at pretest, posttest and 6, 12, 18, and 24 month follow-ups will include indicators of CGM psychological distress (anxiety, depression); CGC adjustment (internalizing and externalizing problems); and disrupted parenting (use of ineffective discipline and low nurturance). Based on the conceptual framework of the prominent Family Stress Model, multi-group structural equation modeling analyses will be used to achieve four aims: (a) To compare the short and long-term effectiveness of CBT and BPT; (b) to examine longitudinally the dynamic linkages between CGM parenting practices, CGM' psychological distress, and CGC adjustment as modified by BPT and CBT; (c) to determine if key moderating variables (race/ethnicity, CGC, initial psychological difficulties in CGC and CGM influence RCT outcomes; and (d) to examine key factors related to acceptability and adherence to the proposed interventions. The findings will inform future clinical practice with custodial grandfamilies by identifying which of the proposed interventions are most effective and most acceptable among specific sub-groups (e.g., race/ethnicity; initial risk) and by unraveling the specific antecedent-consequent relations among CGM distress, dysfunctional parenting, and CGC adjustment.

ELIGIBILITY:
Inclusion Criteria:

* Grandmother raising grandchildren
* No biological resides in grandmother's home
* At least one grandchild between ages 4 and 12
* Grandchild has lived with grandmother for minimum of 3 months
* Grandchild is expected to stay with grandmother

Exclusion Criteria:

* Biological parent is directly involved in raising child
* Grandmother is unable to leave the home to attend weekly meetings
* Grandmother is unable to speak English
* Grandmother is unable to answer simple questions

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in Parenting Quality after intervention up to two years | post-test (2 to 6 weeks following intervention), 6 mos, 12 mos, 18 mos, 2 years
  Parenting quality will be measured in terms of the degree to which grandparents employ positive discipline strategies and engage in warm or nurturing parenting styles. Measured both using self-report and observer ratings.

SECONDARY OUTCOMES:
Change in Grandchild Internalizing and Externalizing Symptoms after intervention up to two years | post-test (2 to 6 weeks following intervention), 6 mos, 12 mos, 18 mos, 24 mos
  Measured through grandmother report, grandchild report, and observer ratings
Change in GM Psychological Distress after intervention up to two years | post-test (2 to 6 weeks following intervention), 6mos, 12 mos, 18 mos, 24 mos
  Grandmother's psychological distressed as defined by anxiety and depression levels (measured both through self report and clinical ratings)
Intervention efficacy | 2 to 6 weeks following intervention
  GM satisfaction with intervention, and comparative impact of interventions vs. control. These variables will be measured at the post-test which will take place between two and 6 weeks following the completion of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Smith, Ed.D., Principal Investigator — Kent State University; Bert Hayslip, Ph.D., Principal Investigator — University of North Texas Health Science Center; Karie Feldman, Ph.D., Study Director — Kent State University
Locations (4):
- United States (4):
  - University of California, San Bernardino, San Bernardino, California
  - University of Maryland Baltimore County, Baltimore, Maryland
  - Kent State University, Kent, Ohio
  - University of North Texas, Denton, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith GC, Hancock GR, Hayslip B. Predictors and moderators of treatment efficacy in reducing custodial grandmothers' psychological distress. Aging Ment Health. 2022 Feb;26(2):250-262. doi: 10.1080/13607863.2020.1857688. Epub 2021 Jan 4. PMID 33393377
- [Derived] Smith GC, Hayslip B, Hancock GR, Strieder FH, Montoro-Rodriguez J. A randomized clinical trial of interventions for improving well-being in custodial grandfamilies. J Fam Psychol. 2018 Sep;32(6):816-827. doi: 10.1037/fam0000457. PMID 30188171